CLINICAL TRIAL: NCT06146985
Title: A Multicohort, Single-Centre, Phase II Trial of the Efficacy and Safety of Famitinib in Combination With Adebrelimab for the Treatment of Advanced Thyroid Cancer
Brief Title: Famitinib in Combination With Adebrelimab for the Treatment of Advanced Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, QIU WEIHUA, Director, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-IIT-FMTN-SHR-1316
Record Dates: First submitted 2023-11-08; First posted 2023-11-27 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Differentiated Thyroid Cancer refractory to standard treatment（DTC） (Experimental): Participants will receive 1200mg Adebrelimab i.v. once every 3 weeks and 20 mg Famitinib orally before or after the meal every day for 3 weeks until PD and/or endurable toxicity appears.
  Interventions: Combination Product: 20 mg Famitinib & 1200 mg Adebrelimab
- Medullary Thyroid Cancer(MTC) (Experimental): Participants will receive 1200mg Adebrelimab i.v. once every 3 weeks and 20 mg Famitinib orally before or after the meal every day for 3 weeks until PD and/or endurable toxicity appears.
  Interventions: Combination Product: 20 mg Famitinib & 1200 mg Adebrelimab
- Anaplastic Thyroid Carcinoma（ATC） (Experimental): Participants will receive 1200mg Adebrelimab i.v. once every 3 weeks and 20 mg Famitinib orally before or after the meal every day for 3 weeks until PD and/or endurable toxicity appears.
  Interventions: Combination Product: 20 mg Famitinib & 1200 mg Adebrelimab

INTERVENTIONS:
Combination Product: 20 mg Famitinib & 1200 mg Adebrelimab — Famitinib is a novel multi-targeted tyrosine kinase inhibitor targeting VEGFR2, PDGFR, and c-kit. Adebrelizumab is a humanised immunoglobulin G4 (IgG4) monoclonal antibody that binds specifically to human PD-L1

SUMMARY:
This is a multi-cohort, open-label, single-centre, Phase 2 study aiming to investigate the efficacy and safety of a regimen using the multi-targeted kinase inhibitor Famitinib in combination with the PD-L1 antibody Adebrelimab for the patients with unresectable locally advanced or metastatic refractory to standard treatment differentiated thyroid cancer (DTC), medullary thyroid carcinoma (MTC) as well as Anaplastic thyroid carcinoma (ATC).

DETAILED DESCRIPTION:
The participants who meet the inclusion criteria will be assigned to different cohorts to be treated. Participants will receive Adebrelimab 1200 mg intravenously once every three weeks (Q3W), together with Famitinib 20 mg orally daily before or after the diet. Participants will be given the regimen of Famitinib in combination with Adebrelimab during the Treatment phase until disease progression or undulated toxicity appears.

ELIGIBILITY:
Inclusion Criteria:

(1)Sign on the informed consent form. (2)Age between 18 to 75 years old. (3)Histologically or cytologically confirmed unresectable locally advanced or metastatic Differentiated Thyroid Cancer (DTC), locally advanced or metastatic Medullary thyroid cancer (MTC), and Anaplastic Thyroid Cancer (ATC).

(4)DTC has progressed after I-131 or thyroid hormone-treating (match any one of the following conditions):

1. At least one measurable lesion loses the ability of Iodine uptake after Iodine radiation treatment.
2. Disease progression occurs for at least one measurable lesion within 12 months after I-131 treatment, even with the ability of Iodine uptake.
3. Cumulative dose of Iodine treatment ≥ 22.2 (GBq); the final treatment should be six months before enrollment. As for the patients who do not belong to the poorly differentiated subtype, their TSH level should be at the inhibitory level from the Screening phase.

(5)Resistance of Lenvatinib and Anlotinib. (6)BRAF V600E, RET mutation does not exist. (7)At least one measurable lesion. According to the RECIST v1.1, the long diameter through Spiral CT scanning should be no less than 10 mm, or the short diameter of the lymphoid should be no less than 15 mm; the confirmed progressed lesion received local treatment can be regarded as a targeted lesion.

(8)ECOG score between 0 to 1. (9)Laboratory examination confirms that the organ functions are enough within 14 days before the first dose:

1. Blood test: WBC≥3.0×109/L；ANC≥1.5×109/L；PLT≥50×109/L；HGB≥90 g/L
2. Liver function: AST≤3.0×ULN；ALT≤3.0×ULN；TBIL<60 μmol/L;
3. Kidney function: Cr≤1.5×ULN or CrCl ≥30 mL/min;
4. Coagulation function: INR≤1.5，APTT≤1.5 ×ULN
5. HBV-DNA≤2×103IU/ml (The participants whose HBV-DNA> 2×103IU/ml should taking anti-virus treatment after enrollment).

(10)Male participants, as well as females of childbearing age, must take contraceptive measures from the start of the first dose to 3 months after the final dose.

Exclusion Criteria:

1. Previous or simultaneous concomitant with other malignant tumors (except treated non-malignant melanoma skin cancer, cervical carcinoma in situ, papillary thyroid cancer).
2. Has been treated by immunotherapy, such as PD-1 antibody, PD-L1 antibody, and CTLA-4 antibody.
3. With the cardiac clinical symptoms or diseases which cannot be controlled well, such as:

1) Class 2 and upper classes of cardiac insufficiency (according to NYHA), or cardiac color ultrasound examination confirms LVEF < 50 %.

2) Unstable Angina Pectoris. 3) Myocardial infarction occurs in one year before research. 4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.

5) Female: QTc>470ms; Male: QTc>450ms. (Calculated by Fridericia formula; average value of 3 tests can be used if QTc shows abnormal results every 2 min).

(4)Previous hypertensive crisis or hypertensive encephalopathy or high blood pressure which cannot be reduced to normal range by antihypertensive medication (systolic blood pressure≥140mmHg or diastolic blood pressure ≥90mmHg). Taking antihypertensive medication is acceptable to achieve the upper parameter.

(5)Have multiple factors affect oral absorption, such as inability to swallow, nausea and vomiting, chronic diarrhea, and intestinal obstruction.

(6)Have risks of gastrointestinal bleeding including:

1. Those who have active peptic ulcer lesions and positive fecal occult blood;
2. Those with a history of melena and hematemesis within 3 months. (7)Abnormal coagulation function (INR>1.5×ULN、APTT>1.5×ULN) or the ones who have the trend of bleeding.

(8)Have a history of organ transplantation or hepatic encephalopathy. (9)Have immunodeficiency disease within 7 days before the first dose, or are receiving systemic hormone therapy (≥10 mg/day prednisone or other hormones at equal doses), or other forms of immunosuppressive therapy.

(10)Severe allergic reaction for Iodinated contrast media, antibody drugs, and anti-angiogenic drugs. (≥ Class 3) (11)Have taken part in other clinical trials or taken other experimental drug within 4 weeks before the first dose.

(12)A positive pregnancy test at baseline in a pregnant or breastfeeding woman or a woman of childbearing age.

(13)Other factors that may affect subject safety or trial compliance as judged by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  ORR was defined as the percentage of participants with the best overall response (BOR) of complete response (CR) or partial response (PR) as measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Disease control rate (DCR) | From date of treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  DCR is defined as the proportion of participants with complete response (CR), partial response (PR) and stable disease (SD) as measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Progression-free survival (PFS) | From date of treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS is defined as the time from the date of randomisation to the date of first documentation of PD or date of death, whichever occurs first, as measured by RECIST V1.1.
Overall Survival (OS) | From date of treatment start until the date of death from any cause, assessed up to 60 months
  OS is defined as the time from treatment to death, regardless of disease recurrence.
Safety Assessment | From treating to the date AEs, SAEs, or abnormal results occurs. assessed up to 60 months
  The safety assessment includes the rate of treatment-related adverse effects, severe adverse effects, and abnormal laboratory examination results, which have clinical significance according to CTCAE v 5.0.